CLINICAL TRIAL: NCT06050174
Title: Efficacy of Locally Delivered Azadirachta Indica (Neem) Extract as an Adjunct to Non-Surgical Periodontal Management
Brief Title: Azadirachta Indica (Neem) Extract as an Adjunct to Non-Surgical Periodontal Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-RECD962
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Periodontitis
Keywords: Periodontitis; Azadirachta Indica; Locally Delivery; TNF-α
MeSH Terms: conditions — Periodontitis | interventions — neem oil; Periodontal Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azadirachta Indica (Experimental): Azadirachta Indica (neem) gel are locally delivered to deepest part of the periodontal pocket by syringe with blunted tip gently and removed slowly in order not to harm the tissue for group 1 patients after phase 1 therapy by two weeks.
  Interventions: Drug: Azadirachta Indica; Procedure: Non Surgical Periodontal Therapy
- Non Surgical Periodontal Therapy (Placebo Comparator): The patients will receive full mouth one stage debridement using ultrasonic scalers, manual scalers and curettes with oral hygiene instructions and education.
  Interventions: Procedure: Non Surgical Periodontal Therapy

INTERVENTIONS:
Drug: Azadirachta Indica — Azadirachtaindica L. is a multipurpose medicinal tree of family Meliaceae.Is also named "Nimba", "holy tree", "Vembu", "Arishtha", "Indian neem tree", "Indian lilac", "wonder tree. It occurs in tropical and semitropical regions of the world. Almost all parts of this incredible tree have been used as phytomedicines for more than 4,000 years.
  Various pharmacological attributes such as antifungal, antiviral, antibacterial, anti-inflammatory, sterilant, antiscabic, antiallergenic and analgesic are attributed to various parts of the tree.
  Other Names: Neem; Nimba; Vembu; Arishtha
  Arms: Azadirachta Indica
Procedure: Non Surgical Periodontal Therapy — The patients will receive full mouth one stage debridement using ultrasonic scalers, manual scalers and curettes with oral hygiene instructions and education.
  Other Names: Periodontal Debridement

SUMMARY:
Azadirachta-Indica has various therapeutic activities such as antiseptic, antiulcer, astringent, superior antiviral and for cleaning the teeth in various dental diseases in vitro and vivo. It also purifies blood, removes toxins from the body and neutralizes free radicals. Due to its therapeutic effects, ease of availability of neem, being cost effective and its safety with no adverse reactions, Azadirachta-Indica has been selected for this study as a local drug delivery in the gel form to be placed in periodontal pockets as an adjunct to non-surgical periodontal debridement for the management of localized periodontitis.

DETAILED DESCRIPTION:
Total number of thirty-two (32) periodontitis patients including both males and females will be included in the study.

To assess the effect of neem gel on the clinical parameters of patients with localized periodontitis t-test or an equivalent non-parametric test will be used for comparison of Intervention group (neem extract gel) and Control group (non-surgical periodontal debridement). At first preoperative periapical radiographs will be taken for assessment of bone level. The patients will receive full mouth one stage debridement using ultrasonic scalers, manual scalers and curettes with oral hygiene instructions and education.

Baseline assessment will be done following phase I therapy by 2 weeks by full mouth periodontal charting and samples from gingival crevicular fluid will be taken using a sterile perio-paper inserted into the deepest periodontal pocket with horizontal bone loss. AzadirachtaIndica Extract Gel will be applied in the deepest pocket by syringe with blunted tip gently and removed slowly in order not to harm the tissue for group 1 patients after phase 1 therapy by two weeks. Follow up of the patients will be done after 3 months after phase I therapy with evaluation of the clinical parameters. The patients will be instructed to brush their teeth 3 times per day during the treatment period using a soft tooth brush together with regular flossing of teeth. A brochure containing written oral hygiene instructions will be given to the patients.

The clinical parameters will be measured two times during the study, the first time at the baseline after two weeks of full mouth debridement and the second time is after baseline by 3 months.

GCF sampling will be done just before neem gel application. Mean values of each parameter will be calculated per patient and per group as well as parameters at the deepest pocket site.

A full mouth periodontal charting will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Both males and females will be included in the age group of 20-55 years old.
2. Patients diagnosed to have (Stage II or Stage III) periodontitis; (3-6 mm CAL, pocket depth ≤ 7 mm, mostly horizontal 15%-33% bone loss as assessed by preoperative radiographs with no tooth loss due to periodontitis).
3. Patients free from systemic diseases according to the modified Burkett's health history questionnaire.
4. Patients who can follow and maintain oral hygiene instructions.
5. Patients who didn't perform any periodontal therapy in the last 6 months.

Exclusion Criteria:

1. Pregnant ladies or lactating mothers.
2. Smokers.
3. Patients with history of allergy against one of the components of neem.
4. Asthmatic patients

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
clinical score | change from baseline at 3 months
  Measuring plaque index, Modified sulcus bleeding index, Probing depth, 4. Clinical attachment level.

SECONDARY OUTCOMES:
Tumor Necrosis Factor alpha | change from baseline at 3 months
  Measuring concentrations of Tumor Necrosis Factor (TNF-α).

CONTACTS AND LOCATIONS:
Overall Officials: Hala A. Abuel-Ela, Professor, Study Director — Faculty of dentistry- Ain shams University
Locations (1):
- Faculty of Dentistry -Ain Shams University, Cairo, Egypt